CLINICAL TRIAL: NCT05705284
Title: The Development and iMplementation Of a Multidisciplinary Medication Review and Deprescribing Intervention Among Frail Older People in primarY Care (MODIFY Study)
Brief Title: MODIFY or Medication Review in Primary Care Study
Acronym: MODIFY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: University of Portsmouth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ERGO ID 71720
Record Dates: First submitted 2022-03-22; First posted 2023-01-30 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Aging
Keywords: polypharmacy

STUDY DESIGN:
Intervention Model Description: Multidisciplinary process for medication review/deprescribing: The intervention will be a structured process for performing a shared-decision, person-centred medication review among those living with frailty involving GPs, PCN-pharmacist and ANPs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients participating in structured multidisciplinary medication review (Experimental): Patients participating in structured multidisciplinary medication review
  Interventions: Other: Structured multidisciplinary medication review

INTERVENTIONS:
Other: Structured multidisciplinary medication review — Multidisciplinary process for medication review/deprescribing: The intervention will be a structured process for performing a shared-decision, person-centred medication review among those living with frailty involving GPs, PCN-pharmacist and ANPs.

SUMMARY:
A third of older people take five or more regular medications (polypharmacy) potentially increasing the risk of side-effects, hospital admission and death, with higher risk among people living with frailty. National recommendations suggest that medications taken by frail older people should be reviewed annually by GPs to identify and reduce/ stop inappropriate medications (deprescribing). Yet this does not happen routinely due to GPs' lack of time, increased workloads and worries about stopping medicines. Recent recommendations suggest involving other non-medical prescribers such as practice-pharmacists and advanced nurse practitioners (ANPs) in reviewing medications. However, it is unknown how staff could work together most effectively and whether they have any training needs.

This research will investigate how practice-pharmacists, ANPs and GPs could best work together with patients living with frailty to perform regular medication reviews. There are four work packages (WPs).

1. Review literature to identify what makes a successful medication review and how to safely deprescribe.
2. Interviews with GPs, practice-pharmacists, ANPs, frail older patients and carers will investigate where medication review should take place, the role of involved parties, type of medications that could be deprescribed, staff training needs, barriers and facilitators for implementation, and strategies to address them.
3. Information from WP1&2 will be used to develop the intervention: a structured medication review process using pharmacists, ANPs and GPs and involving frail patients and their families in decisions about medications. This will be refined through workshops with service users, clinicians and commissioners. A training programme to implement the intervention and increase staff confidence in deprescribing will be developed alongside the intervention.
4. Feasibility study for staff in four GP practices to be trained and to implement the intervention.(this will be subject to further amendment).

DETAILED DESCRIPTION:
Background A third of older people take five or more regular medications (polypharmacy) potentially increasing the risk of side-effects, hospital admission and death. These effects are higher among people living with frailty who lose their in-built reserves and become vulnerable to changes triggered by small events such as a change in medication. National recommendations suggest that medications taken by frail older people should be reviewed annually by their GPs to identify and reduce/ stop inappropriate medications (deprescribing). Yet this does not happen routinely due to GPs' lack of time, increased workloads and worries about stopping medicines.

Recent recommendations suggest involving other non-medical prescribers such as practice-pharmacists and advanced nurse practitioners (ANPs) in reviewing medications. However, it is unknown how staff could work together most effectively and whether they have any training needs.

Aim This research will investigate how practice-pharmacists, ANPs and GPs could best work together with patients living with frailty to perform regular medication review.

Methods The study involves four work packages (WPs). The research team will review previous literature to identify what makes a successful medication review and how to safely reduce/ stop inappropriate medications (WP1).

Interviews with GPs, practice-pharmacists, ANPs, frail older patients and carers will be conducted (WP2). These will discover views about where medication review should take place, the role of each of the involved parties in the process, type of medications that could be deprescribed, staff development and training needs, barriers and facilitators for implementation, and strategies to address these barriers.

Information gathered from WP1&2 will be used to develop the intervention: a structured medication review process using pharmacists, ANPs and GPs most effectively and involving frail patients and their families in decisions about medications (WP3). The intervention will be refined further through a series of workshops with service users, clinicians and commissioners. A training programme to implement the intervention and increase staff confidence in reducing/ stopping medications safely will be developed and delivered to GPs, practice-pharmacists and ANPs based on the Polypharmacy Action Learning Sets approach adopted by the Wessex Academic Health Science Network (AHSN) .

Finally, the feasibility and acceptability of the intervention to staff and patients in four GP practices will be assessed (WP4).

Patient and Public Involvement (PPI) Three PPI members have been involved in protocol development and refinement and will continue to contribute to the research study by for example being involved in developing research instruments and monitoring recruitment.

Dissemination and impact Working with colleagues in the Wessex AHSN and local clinical commissioners, the research team will be able to share our findings and training programme to the wider research and clinical community in Wessex and potentially influence practices and policies both locally and nationally.

ELIGIBILITY:
Eligibility criteria for WP2

Patients:

Inclusion criteria

* Aged 65 and over
* Frail, (as judged by their health care professional, if applicable)
* Prescribed multiple medications (10+), as determined by their health care professional
* Able to give informed consent

Exclusion criteria

* Aged under 65
* Severe cognitive impairment, as judged by their health care professional

Informal carers/ relatives eligibility criteria

Inclusion criteria

* An informal carer/ relative of a frail patient (aged 65 and over) who is taking multiple medications, as identified by a health care professional
* An informal carer/ relative of a patient (aged 65 and over) living with severe dementia who is taking multiple medications, as identified by a health care professional
* Able to consent

Health care professional eligibility criteria

• A health care professional based in GP surgeries in Wessex (eg. GPs, practice-pharmacists, advanced nurse prescriber (ANPs) who works with older people living with frailty, who are prescribed multiple medications.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | Baseline
  proportion of staff recruited and trained in each GP practice
Number of medications | change in scores between baseline and 3 months follow up
  Total number of medications taken by each patient
Rates of adverse events | at 3 months
  rates of adverse drug events due to deprescribing (including self-reported dizziness, falls, drowsiness, confusion, hallucinations, blurred vision, constipation, diarrhoea, dry mouth or other) during 3 months follow up.
Rates of hospitalisation | 3 months
  rates of hospitalisation 3 months post intervention
Mortality rates | 3 months
  mortality rates 3 months post intervention
frailty status | changes between baseline and 3 months
  Frailty score using the electronic frailty index (e-FI)
rates of falls | changes between baseline and 3 months
  number of falls reported and proportion of fallers (self-reported)
Rates of fractures | changes between baseline and 3 months
  number of fractures and proportion of people sustained fractures (self-reported)
function | changes between baseline and 3 months
  Activity of daily living using Barthel
cognition | changes between baseline and 3 months
  - cognition using the abbreviated mental test (AMT)
depression | changes between baseline and 3 months
  - depression using the geriatric depression scale (GDS)
healthcare utilisation | at 3 months follow up
  number of visits to GP/specialists and number of unplanned hospitalisations
Acceptability | at 3 months follow up
  Interviews or focus groups will be conducted at the end of the feasibility study with a purposive sample of (n=6-8) GPs, pharmacists, ANPs in the four GP practices who received the training and implemented the intervention, and 8-10 patients and carers who received the intervention
Feasibility of deprescribing | 3 months follow up
  number of recommendations in the medication reviews made to each patient (stop, reduce, switch or start).
number of potentially inappropriate medications | Change between baseline and 3 months follow up
  total number of potentially inappropriate medications months using the STOPP/START criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Kinda Ibrahim, PhD, Principal Investigator — University of Southampton
Locations (1):
- Clinical Research Network in Primary Care, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The development and iMplementation Of a multidisciplinary medication review and Deprescribing Intervention among Frail older people in primarY care — https://www.arc-wx.nihr.ac.uk/research-areas-list/modify%3A-the-development-and-implementation-of-a-multidisciplinary-medication-review-and-deprescribing-intervention-among-frail-older-people-in-primary-care